CLINICAL TRIAL: NCT06097260
Title: A Randomized, Double-blind, Dose-ranging, Placebo-controlled Study to Evaluate the Efficacy and Safety of Bexotegrast (PLN-74809) for the Treatment of Idiopathic Pulmonary Fibrosis (BEACON-IPF)
Brief Title: Randomized, Double-blind Study of Efficacy and Safety of Bexotegrast (PLN-74809) for Idiopathic Pulmonary Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMB recommendation
Sponsor: Pliant Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLN-74809-IPF-206; BEACON-IPF (Other: Pliant Therapeutics Inc)
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: IPF; idiopathic pulmonary fibrosis; pulmonary fibrosis; bexotegrast; Beacon; BEACON-IPF
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Experimental): Placebo
  Interventions: Drug: Placebo
- Bexotegrast (PLN-74809) 160 mg Dose (Experimental): Bexotegrast (PLN-74809) 160 mg Dose - 52 weeks
  Interventions: Drug: PLN-74809
- Bexotegrast (PLN-74809) 320 mg Dose (Experimental): Bexotegrast (PLN-74809) 320 mg Dose - 52 weeks
  Interventions: Drug: PLN-74809

INTERVENTIONS:
Drug: PLN-74809 — PLN-74809
  Arms: Bexotegrast (PLN-74809) 160 mg Dose; Bexotegrast (PLN-74809) 320 mg Dose
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A randomized, double-blind, dose-ranging, placebo-controlled study to evaluate the efficacy and safety of bexotegrast (PLN-74809) for the treatment of idiopathic pulmonary fibrosis (BEACON-IPF).

DETAILED DESCRIPTION:
This is a randomized, double-blind, dose-ranging, placebo-controlled study to evaluate the efficacy and safety of 2 doses of bexotegrast (PLN-74809) [160 and 320 mg] taken for 52 weeks by participants with IPF taking and not taking background therapy (ie, nintedanib or pirfenidone).

The study will consist of an up to 35-day Screening Period, a 52-week Treatment Period, and a 14 day Safety Follow-up Period. Of note, participants who are not taking background therapy at study entry will be allowed to initiate it at any time during the study.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 40 years of age prior to screening
2. IPF diagnosis ≤ 7 years prior to screening
3. FVCpp ≥ 45%
4. Diffusing capacity for carbon monoxide percent predicted (hemoglobin-adjusted) ≥ 30% and < 90%
5. Current treatment for IPF with background therapy is allowed, if at a stable dose for ≥ 12 weeks prior to screening
6. If not currently receiving treatment for IPF (either treatment naïve or discontinued prior treatment), participant must not have taken background therapy for at least 8 weeks prior to screening

Exclusion Criteria:

1. Receiving pharmacologic therapy for pulmonary hypertension
2. Self-reported smoking of any kind (not limited to tobacco)
3. History of malignancy within the past 5 years or ongoing malignancy other than basal cell carcinoma, resected noninvasive cutaneous squamous cell carcinoma, or treated cervical carcinoma in situ
4. Hepatic impairment or end-stage liver disease
5. Renal impairment or end-stage kidney disease requiring dialysis
6. Pregnant or lactating female participant
7. Uncontrolled systemic arterial hypertension
8. Receiving any unapproved or investigational agent intended for treatment of fibrosis in IPF
9. Prior administration of bexotegrast
10. Likely to have lung transplantation during the study (being on transplantation list is not an exclusion)
11. Forced expiratory volume in the first second (FEV1)/FVC ratio <0.7 at screening
12. Clinical evidence of active infection, including, but not limited to bronchitis, pneumonia, or sinusitis that can affect FVC measurement during screening or at randomization
13. Known acute IPF exacerbation, or suspicion by the Investigator of such, 6 months prior to screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
To characterize the effect of bexotegrast versus placebo on the change in forced vital capacity (FVC) in participants with idiopathic pulmonary fibrosis (IPF) | 52 weeks
  Change from baseline in absolute FVC (mL) at Week 52

SECONDARY OUTCOMES:
To characterize the effect of bexotegrast versus placebo over 52 weeks of treatment on disease progression | Up to 52 weeks
  • Time to disease progression, defined as time to first occurrence of ≥10% absolute decline from baseline in forced vital capacity percent predicted (FVCpp), adjudicated respiratory-related hospitalization, adjudicated acute IPF exacerbation or all-cause mortality through Week 52
Time to disease progression defined as | Up to 52 weeks
  Time to first occurrence of adjudicated respiratory-related hospitalization, adjudicated acute IPF exacerbation or all-cause mortality through Week 52
Proportion of participants with disease progression defined as | Up to 52 weeks
  Proportion of participants with a ≥10% absolute decline in FVCpp from baseline or all-cause mortality through Week 52
To characterize the effect of bexotegrast versus placebo on the change in FVC in participants with and without background therapy at baseline with IPF | 52 weeks
  Change from baseline in absolute FVC (mL) at Week 52
  * In participants on background therapy at baseline
  * In participants not on background therapy at baseline
Change from baseline in Living with Pulmonary Fibrosis (L-PF) Dyspnoea and Cough Domain score | 52 Weeks
  The Living with Pulmonary Fibrosis (L-PF) questionnaire assesses symptoms and quality of life in patients with fibrosing interstitial lung diseases (ILDs). Its Dyspnoea and Cough domains, whose items' responses are based on a 24-hour recall, have scores ranging from 0 to 100, with higher scores indicating greater symptom severity. Domain and total scores range from 0 to 100, with higher scores indicating greater impairment.
Change from baseline in King's Brief Interstitial Lung Disease (K-BILD) questionnaire Total score | 52 Weeks
  The KBILD(King's Brief Interstitial Lung Disease Questionnaire) is a self-completed health status questionnaire that comprises 15 items and a seven-point Likert response scale.1 It has three domains: psychological, breathlessness and activities and chest symptoms. The KBILD domain and total score ranges are 0-100; 100 represents best health status
To characterize the effect of bexotegrast versus placebo on change in lung fibrosis by high-resolution computed tomography | 52 Weeks
  Absolute change from baseline in quantitative lung fibrosis (QLF) extent (%)
To characterize the safety and tolerability of bexotegrast versus placebo in participants with IPF | Up to 52 weeks
  Proportion of participants with treatment-emergent adverse events and serious adverse events
To characterize the safety and tolerability of bexotegrast versus placebo in participants with IPF over 52 weeks of treatment | Over 52 Weeks
  Number of participants with Adverse Events (AEs) Number of participants with Serious AEs (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Pliant Therapeutics Medical Monitor, Study Director — Pliant Therapeutics, Inc.
Locations (267):
- United States (79):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - Dignity Health-St. Josephs Hospital and Medical Center, Phoenix, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Newport Native MD, Inc, Newport Beach, California
  - Palmtree Clinical Research, Palm Springs, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Paradigm Clinical Research Institute Inc - ClinEdge, Redding, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center - Pulmonary Practice, San Francisco, California
  - Jeffrey S. Sager, MD Medical Corporation, Santa Barbara, California
  - Stanford Health Care, Stanford, California
  - University of Colorado, Aurora, Colorado
  - National Jewish Health Main Campus, Denver, Colorado
  - Critical Care, Pulmonary and Sleep Associates, Lakewood, Colorado
  - Nuvance Health Medical Practices, Pulmonary & Sleep Specialists, Danbury, Connecticut
  - Yale New Haven Hospital - York Street Campus, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Clinical Research Specialists, LLC, Kissimmee, Florida
  - Clinical Site Partners - Leesburg, Leesburg, Florida
  - Central Florida Pulmonary Group PA, Orlando, Florida
  - GCP Clinical Research, Tampa, Florida
  - Emory Clinic, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - IU Health Advanced Heart and Lung Care, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Lexington VA Medical Center, Lexington, Kentucky
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - The Johns Hopkins Hospital JHH, Baltimore, Maryland
  - Massachusetts General Hospital - Pulmonary Associates, Boston, Massachusetts
  - Brigham and Womans Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Cente, Boston, Massachusetts
  - Infinity Medical Research, North Dartmouth, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - The Lung Research Center, Chesterfield, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - New York Presbyterian Hospital-Columbia University Medical Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Montefiore Medical Center Moses Division Hospital, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - PulmonIx, LLC, Greensboro, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - OU Health Physicians, Oklahoma City, Oklahoma
  - Bend Memorial Clinic/Summit Medical Group - Eastside, Bend, Oregon
  - Legacy Good Samaritan Hospital, Portland, Oregon
  - Clinical Research Associates Of Central PA , LLC, DuBois, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Velocity Clinical Research, Greenville, South Carolina
  - Lowcountry Lung and Critical Care PA, North Charleston, South Carolina
  - Clinical Trials Center of Middle Tennessee, Franklin, Tennessee
  - Statcare Pulmonary Consultants - Knoxville, Knoxville, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott and White Health - Advanced Lung Disease Specialists, Dallas, Texas
  - El Paso Pulmonary Association, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas
  - Research Centers of America, McKinney, Texas
  - Renovatio Clinical Research, The Woodlands, Texas
  - Topline Clinical Research, Waxahachie, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - INOVA Fairfax Medical Campus, Falls Church, Virginia
  - Western Washington Medical Group, Everett, Washington
- Argentina (16):
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - Instituto Ave Pulmo, Mar del Plata, Buenos Aires
  - Clinica Privada Independencia, Munro, Buenos Aires
  - Centro Respiratorio Quilmes, Quilmes, Buenos Aires
  - CEMER - Centro Medico de Enfermedades Respiratorias, Vicente López, Buenos Aires
  - Centro de Investigacion Clinica-CEDIC, Buenos Aires, Ciudad Autonoma Buenos Aires
  - Centro Médico Dra de Salvo, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Instituto Medico Fundacion Grupo Colaborativo Rosario Investigacion y Prevencion Medica, Rosario, Santa Fe Province
  - Instituto Médico de la Fundación Estudios Clínicos, Rosario, Santa Fe Province
  - Sanatorio Parque de Rosario, Rosario, Santa Fe Province
  - Centro Integral de Medicina Respiratoria (CIMER), San Miguel de Tucumán, Tucumán Province
  - Consultorios Médicos Organización de Buen Ayre SRL, Buenos Aires
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Instituto de Medicina Respiratoria, Córdoba
  - Fundacion Scherbovsky, Mendoza
  - INSARES, Mendoza
- Australia (11):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Lung Research Qld, Chermside, Queensland
  - Respiratory Clinical Trials, Kent Town, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - TrialsWest, Spearwood, Western Australia
  - Institute for Respiratory Health - Midland, Midland
- Belgium (2):
  - AZ Delta, Roeselare, West-Vlaanderen
  - UZ Leuvan, Leuven
- Brazil (8):
  - Hospital Cardio Pulmonar, Salvador, Estado de Bahia
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Instituto Mederi de Pesquisa e Saude, Passo Fundo, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre HCPA - PPDS, Porto Alegre
  - Hospital São Lucas da PUCRS, Porto Alegre
- Canada (5):
  - Kelowna Respirology and Allergy Research, Kelowna, British Columbia
  - Pacific Lung Research Center, Vancouver, British Columbia
  - Dynamic Drug Advancement, Ajax, Ontario
  - CIC Joliette, Saint-Charles-Borromée, Quebec
  - Centre d'investigation Clinique Mauricie, Trois-Rivières, Quebec
- Chile (6):
  - CENRESIN, Quillota
  - Av. Providencia 1208 oficina 209, Santiago
  - CIMER - Centro de Investigaciones Medicas Respiratorias, Santiago
  - CEC SpA, Santiago
  - Biocinetic, Santiago
  - Centro de Investigacion del Maule, Talca
- China (17):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The 3rd Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial Chest Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Yichang Central People's Hospital, Yichang, Hubei
  - The second Xiangya Hospital of Central South University, Changsha, Hunan
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Academy of Medical Sciences · Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
- Czechia (3):
  - Fakultni Nemocnice Olomouc, Olomouc, Olomoucký kraj
  - Fakultni nemocnice Brno, Brno, South Moravian
  - Fakultni Thomayerova Nemocnice, Prague
- Denmark (4):
  - Odense Universitetshospital, Odense, Region Syddanmark
  - Aarhus Universitetshospital, Aarhus
  - Gentofte Hospital, Hellerup
  - Odense Universitetshospital, Odense
- France (14):
  - Hôpital Pontchaillou, Rennes, Ille-et-Vilaine
  - Institut Coeur Poumon - CHU de Lille, Lille, Nord
  - Hôpital Avicenne, Bobigny, Seine Saint Denis
  - CHU de Bordeaux- Hopital du Haut Lévêque, Bordeaux
  - CHU Lyon - Hôpital Cardio-Vasculaire et Pneumologique Louis Pradel, Lyon
  - Hôpital Nord - CHU Marseille, Marseille
  - CHU Arnaud de Villeneuve, Montpellier
  - CHU Nice - Hôpital Pasteur, Nice
  - Hopital Pasteur CHU Nice, Nice
  - Hospital Bretonneau, Paris
  - Hôpital Bichat - Claude Bernard, Paris
  - Hopital Haut-Leveque Pharmacie, Pessac
  - CHU Reims - Hôpital Maison Blanche, Reims
  - Hopital Larrey, Toulouse
- Germany (10):
  - LMU Klinikum der Universität München - Campus Großhadern, München, Bavaria
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Kliniken der Stadt Koln, Cologne, North Rhine-Westphalia
  - Ruhrlandklinik, Essen, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein
  - Evangelische Lungenklinik Berlin, Berlin
  - Fachkrankenhaus Coswig GmbH, Coswig
  - IKF Pneumologie GmbH & Co. KG, Frankfurt
  - Universitaetsklinikum des Saarlandes, Homburg
  - Universitaetsklinikum Leipzig AoeR, Leipzig
- Greece (4):
  - University General Hospital of Patras, Pátrai, Achaïa
  - Sotiria Thoracic Diseases Hospital of Athens, Athens, Attica
  - University General Hospital of Alexandroupolis, Alexandroupoli, Evros
  - University General Hospital of Heraklion, Heraklion
- India (11):
  - Unity Hospital ICU and Trauma, Surat, Gujarat
  - ESIC Medical College and Hospital, Faridabad, Haryana
  - K.L.E. Society's Dr. Prabhakar Kore Hospital and Medical Research Centre, Belagavi, Karnataka
  - BHS Lakeview Hospital, Belagavi, Karnataka
  - Bhatia Hospital, Mumbai, Maharashtra
  - Siddhi Hospital, Nashik, Maharashtra
  - J.L.N., Medical College and Attached Hospitals, Ajmer, Rajasthan
  - Asthma Bhavan, Jaipur, Rajasthan
  - Midland Healthcare & Research Center, Lucknow, Uttar Pradesh
  - Calcutta Medical Research Institute, Kolkata, West Bengal
  - B. P. Poddar Hospital and Medical Research Limited, Kolkata, West Bengal
- Israel (10):
  - Kaplan Medical Center, Rehovot, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Barzilai Medical Center, Ashkelon, Southern District
  - Tel Aviv Sourasky Medical Center, Ashkelon, Tel Aviv
  - Sheba Medical Center, Ramat Gan, Tel Aviv
  - Soroka University Medical Center, Beersheba
  - Lady Davis Carmel Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
- Italy (5):
  - Ospedale San Giuseppe Multimedica SpA, Milan, Milano
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - ASST Papa Giovanni XXIII - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti di Foggia, Foggia
- Japan (23):
  - NHO Kyushu Medical Center, Fukuoka, Fukuoka
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Aso Co.,Ltd Iizuka Hospital, Iizuka-shi, Fukuoka
  - Hospital of the University of Occupational and Environmental Health, Kitakyushu-shi, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Hiroshima Prefectural Hospital, Hiroshima, Hiroshima
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kobe City Hospital Organization, Kobe, Hyōgo
  - Center General Hospital, Kobe, Hyōgo
  - NHO Ibarakihigashi National Hospital, Naka-gun, Ibaraki
  - Tokushima University Hospital, Kawasaki-shi, Kanagawa
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Okayama University Hospital, Okayama, Okayama-ken
  - NHO Kinki-Chuo Chest Medical Center, Osaka, Osaka
  - Saitama Prefectural Cardiovascular and Respiratory Center, Kumagaya-shi, Saitama
  - Saitama Red Cross Hospital, Saitama-shi, Saitama
  - Shimane University Hospital, Izumo-shi, Shimane
  - Hamamatsu University School of Medicine, University Hospital, Hamamatsu, Shizuoka
  - Institute of Science Tokyo Hospital, Bunkyō City, Tokyo-To
  - Nippon Medical School Hospital, Bunkyō City, Tokyo-To
  - NHO Okinawa National Hospital, Hachioji-shi, Tokyo-To
  - Juntendo University Hospital, Minatoku, Tokyo-To
- Netherlands (2):
  - VU Medisch Centrum, Amsterdam, North Holland
  - St. Antonius Ziekenhuis, Nieuwegein, Utrecht
- New Zealand (4):
  - Christchurch Hospital, Christchurch, Canterbury
  - Greenlane Clinical Centre, Auckland, North Island
  - Dunedin Hospital, Dunedin, Otago
  - Waikato Hospital, Hamilton, Waikato Region
- Poland (4):
  - Twoja Przychodnia NCM, Nowa Sól, Lubusz Voivodeship
  - Vitamed Galaj i Cichomski sp.j., Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
- Portugal (3):
  - Hospital de Braga, Braga
  - Centro Hospitalar de Lisboa Central, E.P.E - Hospital de Santa Marta, Lisbon
  - Centro Hospitalar Vila Nova de Gaia/Espinho, E.P.E., Vila Nova de Gaia
- South Korea (6):
  - Inje University Busan Paik Hospital, Pusan, Gyeongsangnam-do
  - Korea University Anam Hospital, Seoul, Seoul Teugbyeolsi
  - Hanyang University Medical Center, Seoul, Seoul Teugbyeolsi
  - Inje University Haeundae Paik Hospital, Busan
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (5):
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - CHUS - H. Clinico U. de Santiago, Santiago de Compostela
- Taiwan (6):
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei
- United Kingdom (9):
  - Royal Papworth Hospital, Cambridge, Cambridgeshire
  - Peterborough City Hospital, Peterborough, Cambridgeshire
  - Altnagelvin Area Hospital, Londonderry, Derry
  - Southampton General Hospital, Southampton, Hampshire
  - Castle Hill Hospital, Cottingham, North Humberside
  - Churchill Hospital, Oxford, Oxfordshire
  - Pinderfields General Hospital, Wakefield, West Yorkshire
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Trial website — https://www.beaconipf.com/